CLINICAL TRIAL: NCT06895057
Title: Comparison of the Effects of Telerehabilitation and Clinic-Applied Core Stabilization Exercises on Pain, Quality of Life and Endurance in Patients With Chronic Low Back Pain
Brief Title: Telerehabilitation and Clinic-Applied Core Stabilization Exercises in Patients With Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Zekiye Beyza Kolukısa, physiotherapist, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIBTU-FTR--ZBK-1
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Low Back Pain, Chronic
Keywords: Chronic low back pain, exercise, telerehabilitation, core stabilization
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telerehabilitation group (Experimental): The exercise program will be applied online via tablet.Individuals who will participate in the study will be put into practice twice a week for 8 weeks, each session lasting 50 minutes. Pain, quality of life, endurance, functionality, and flexibility assessments will be taken face to face before and after the application for both groups. The treatment satisfaction scale (PGIC) will be taken from both groups in the 4th and 8th weeks. All assessments will be made face to face by the same therapist in the clinic, twice before and after the training.
  The core stabilization exercise program to be applied is planned as follows.
  * Warm-up exercises (10 minutes) (Straight leg raise, circle drawing, side opening)
  * Finding neutral spine position (Pelvic Tilt)
  * Bridge exercise, (one leg pull-up in bridge, bridge rise, fixed hold)
  * Table (abdominal exercise)
  * Crawling position stretching exercises
  * Plank exercises (Advanced plank exercises such as fixed hold, side plank, single leg pull-up
  Interventions: Other: Exercise
- clinical practice group (Experimental): The exercises will be applied face to face to the clinical practice group. Individuals who will participate in the study will be put into practice twice a week for 8 weeks, each session lasting 50 minutes. Pain, quality of life, endurance, functionality, and flexibility assessments will be taken face to face before and after the application for both groups. The treatment satisfaction scale (PGIC) will be taken from both groups in the 4th and 8th weeks. All assessments will be made face to face by the same therapist in the clinic, twice before and after the training.
  The core stabilization exercise program to be applied is planned as follows.
  * Warm-up exercises (10 minutes) (Straight leg raise, circle drawing, side opening)
  * Finding neutral spine position (Pelvic Tilt
  * Bridge exercise, (one leg pull-up in bridge, bridge rise, fixed hold)
  * Table (abdominal exercise)
  * Crawling position stretching exercises
  * Plank exercises (Advanced plank exercises such as fixed hold, side plank
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Individuals who voluntarily accept to participate in the study will be divided into two groups as telerehabilitation and clinical practice groups by randomization. Exercises will be applied face to face to the clinical practice group and online to the telerehabilitation group via tablet. Individuals who will participate in the study will be applied twice a week for 8 weeks, each session lasting 50 minutes. Pain, quality of life, endurance, functionality, and flexibility assessments will be taken face to face for both groups before and after the application. Treatment satisfaction scale (PGIC) will be taken from both groups in the 4th and 8th weeks. All assessments will be evaluated twice before and after the training by the same therapist in the clinic, face to face.

SUMMARY:
The aim of the study is to compare the effects of core stabilization exercises on pain, quality of life and endurance in individuals with chronic low back pain with telerehabilitation and in-clinic application. In this way, the effect of low-cost, easy-to-access and longer-term telerehabilitation in the treatment of chronic low back pain will be examined comparatively with face-to-face application.

DETAILED DESCRIPTION:
Low back pain is a common health problem worldwide, characterized by the persistence of its symptoms. It usually occurs as a musculoskeletal injury that can occur at work, during exercise, after a traumatic event, or from a condition of unknown cause. According to the National Institutes of Health, 80% of adults experience low back pain in their lifetime. Data from the 2015 National Health Interview Survey showed that the population with low back pain is over 140 million annually. Nonspecific low back pain is a type of pain where the cause cannot be specifically determined, such as tumors, spinal fractures, or infections. According to its duration, low back pain is classified as: acute pain (lasting less than 6 weeks); subacute pain (lasting between 6 weeks and 3 months); or chronic pain (lasting longer than 3 months).

There are various methods for the treatment of chronic low back pain. The aim of the treatment methods is to reduce pain, increase functionality and prevent deterioration in daily life activities. There is strong evidence in treatment-oriented studies that exercise training reduces pain and improves quality of life. The core region is responsible for the transfer of power between the upper and lower extremities of the body. All movements start from the core region and are transferred to the extremities. It is also the most important muscle group that provides body stabilization. The stability of the spine is negatively affected in people with low back pain. Generally, individuals with pain problems have poorly coordinated muscles around the spine and weakness in the core region. Core stabilization exercises aim to improve the strength and control of the muscles that are central to maintaining spinal stability. Telerehabilitation is an online or offline tool that allows personalized treatment of patients. It also allows patients to access information about their treatment and condition at any time. This reduces costs and geographical barriers. The aim of the study is to compare the effects of core stabilization exercises on pain, quality of life and endurance in individuals with chronic low back pain with telerehabilitation and in-clinic application. In this way, the effect of low-cost, easy-to-access and longer-term telerehabilitation in the treatment of chronic low back pain will be examined comparatively with face-to-face application.

ELIGIBILITY:
Inclusion Criteria:

* People with chronic back pain between the ages of 25-55
* People with back pain for more than 3 months
* Ability to read and understand Turkish
* Volunteer to participate in the study
* Those with pain intensity above 3 on the Visual Analog Scale (VAS)

Exclusion Criteria:

* Not accepting to participate in the study,
* Having any pathology that causes back pain (e.g. infections, tumors or rheumatoid arthritis)
* Having liver, heart, lung, kidney failure or tumor
* Having a history of cerebrovascular disease
* Having a neurological disease or skeletal muscle degenerative disease
* Using assistive devices
* Having cognitive disorders
* Being pregnant
* Having undergone orthopedic surgery in the last two years
* Those with scoliosis

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | At Baseline and 8 weeks after the baseline
  The Visual Analog Scale (VAS) will be used to digitize some data that cannot be measured numerically. VAS, developed by Max Freyd, is the most commonly used measurement method in the assessment of pain. The two extreme definitions of the parameter to be evaluated are written on the scale at both ends of a 100-millimeter line, and the patient is asked to indicate by marking the appropriate place on this line for his/her own situation. The starting point of the scale represents no pain, and the ending point represents the most severe pain.
Quality of Life Scale Short Form (SF-36) | At Baseline and 8 weeks after the baseline
  This scale is one of the most common measures used to measure quality of life. It is a questionnaire that examines 8 parameters of health such as physical function, social function, mental health, vitality (energy), pain, role limitations (due to physical and emotional problems), and general perception of health with 36 items. The scale is a self-assessment scale. It can be completed in a short time. Instead of obtaining a single score at the end of the scale, each parameter has its own scoring. A score of 0 indicates poor health status, while 100 indicates good health status. Questions 3-12 are used for physical function, 13-16 for physical role difficulty, 17-19 for emotional role difficulty, 23,27,29,31 for energy, 24,25,26,28,30 for mental health, 20 and 32 for social functioning, 21-22 for pain, and 1 and 33-36 for general perception of health. Each item is scored mathematically according to the answer given within itself. For example, for emotional role difficulty, the transform
Mcgill Body Endurance Tests | At Baseline and 8 weeks after the baseline
  Trunk flexion test: Individuals will be positioned with the soles of their feet on the floor, with knees and hips at 90° flexion, trunk at 60° flexion, and hands crossed on both shoulders. All individuals will be asked to maintain this position and a chronometer will be used to measure at the same time. When the position is disrupted, the test will be terminated and the elapsed time will be recorded in seconds. Trunk extension test: Individuals will be assessed in the prone position. Individuals will be asked to hang from the bed starting from the spina iliaca anterior superior and arms will be crossed on both shoulders. The lower extremity will be fixed by the researcher and individuals will be asked to move their trunks backwards. Trunk lateral bridge test: Individuals will be evaluated on both the right and left sides. For the right side, individuals will be positioned on the forearm with the arm perpendicular to the body, with the elbow flexed at 90°, with the body facing forward.
Oswestry Scale | At Baseline and 8 weeks after the baseline
  The purpose of this index is to measure the functionality levels of individuals with low back pain. It evaluates the changes in parameters such as patients' lifting, pain intensity, personal care, sitting, walking, standing, traveling, social life, and sleeping when they are in pain. There are 6 propositions under each parameter. Patients choose the most appropriate proposition for them. In this way, a total score is obtained by obtaining a score between 0-5 from each question. A maximum of 50 points can be obtained as a result of the test. The score received by the patient is divided by the maximum score that can be obtained, which is 50, and the result obtained is multiplied by 100 to obtain the patient's score from the index.
Modified Schober Test | At Baseline and 8 weeks after the baseline
  It will be used to evaluate the flexibility of the individuals to be included in the study. Both posterior spina iliaca will be marked. 10 cm above and 5 cm below the marked area is determined, the individual is asked to bend forward, the difference between the initial value will be recorded in cm. This measurement will be made to the patient twice, at the beginning of the treatment and at the end of the treatment. A difference of 0-5 cm in the test indicates that flexion flexibility has decreased, while a difference of over 10 cm indicates that flexibility has increased. Values between 5-10 cm are considered normal.
Patient Global Indicator of Change (PGIC) | At Baseline, 4 and 8 weeks after the baseline
  It will be used as a scale of recovery and satisfaction in the 4th and 8th weeks of treatment. It is a 7-point scale that reflects the patient's evaluation of the effectiveness of the treatment. 1=No change, 2=Almost the same, 3=Slightly better, 4=Slightly better, 5=Moderately better, 6=Better, 7=Much better

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Islam Science and Technology University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No